CLINICAL TRIAL: NCT03899896
Title: Voice Feminisation in Transgender Women
Acronym: FemVoc
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Speech Therapy; Transgender Women; Gender Dysphoria
MeSH Terms: conditions — Communication Disorders; Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The voice is a reflection of our identity. In the case of transgender women, there may be a gap between perceived male voice and female appearance. Indeed, hormonal treatment in transgender women has no effect on the voice quality. This gap can have negative consequences on everyday life in banal situations such as telephonic contact leading to limited use of phone calls and social isolation.

Differences between female and male voices seem to be socially determined and do not depend directly on sexual dimorphism of the phonatory organs.

Speech therapy might thus be indicated as a vocal support for transgender women.

Only few studies have examined the impact of perceived voice on the quality of life of transgender women.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Follow-up in the Department of Endocrinology, Diabetology and Nutrition of the University Hospital of Nancy
* Gender dysphoria according to the ICD 11
* Voluntary, informed consent to participate in research
* Compulsory affiliation to the social security system

Exclusion Criteria:

-Refusal or incapacity to be involved in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation to the study will be proposed consecutively to all subjects, fulfilling inclusion criteria, attending in-office follow-up visit for gender dysphoria in the Department of Endocrinology, Diabetology and Nutrition of the University Hospital of Nancy
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
To measure the perceptions of transgender women regarding their voice | 1 year
  Transsexual voice questionnaire Male-to-Female Transsexuals (Dacakis G et al J Voice, 2017): the questionnaire evaluates voice perception in 6 domains: 1 / effect of voice on ease of social interactions, 2 / effect of voice on emotions; 3 / relationship between voice and gender identity, 4 / effort and concentration required to produce voice; 5 / physical aspects of voice production; 6 / pitch. The questionnaire has 30 items. The subject indicates on a 4-point Likert scale ranging from "never or rarely" to "often enough or all the time", the frequency with which he usually feels the symptoms listed. The score is calculated from a minimum of 30 points to a maximum of 120 points

SECONDARY OUTCOMES:
generic quality of life: physical functioning, limitations due to physical state, pain, mental health, limitations due to mental state, social health, vitality and global health | 1 year
  Questionnaire (Short form 36 health survey) The SF-36 is a generic quality of life self-questionnaire with 36 items grouped in 8 dimensions (physical functioning, limitations due to physical state, pain, mental health, limitations due to mental state, social health, vitality and global health). For each dimension a quality of life score is calculated and normalized between 0 (worst possible QoL) and 100 (best QoL possible).
Anxiety: State-Trait Anxiety Inventory, STAI-Y | 1 year
  * The STAI-Y assesses anxiety as a personality trait and as a specific emotional response to a situation. The first part, STAI-Y-1, consists of 20 sentences assessing the current emotional state of the subject. The second part, STAI-Y-2, consists of 20 sentences assessing the subject's usual emotional state.
  * Each answer to an item in the STAI-Y is scored from 1 to 4, with 1 indicating the lowest degree of anxiety and 4 the highest degree of anxiety.
  * In the STAI-Y-1, the subject indicates the intensity of his feelings on a 4-point Likert scale ranging from "not at all" to "many". In the STAI-Y-2, the subject indicates on a 4-point Likert scale ranging from "almost never" to "almost always", a frequency at which he usually feels the symptoms listed.
  * To obtain the score for the STAI-Y-1, the scores for the 20 items (1 to 20) are summed. To obtain the STAI-Y-2 score, the scores for the 20 items (21 to 40) are summed. Each score can therefore vary from 20 to 80.
Self-esteem : Physical self inventory, 25 items (PSI-25) | 1 year
  * The PSI-25 is an inventory of self-esteem relating to the body domain.
  * This tool consists of 6 scales: at the general level, the overall self-esteem scale, at the physical domain level:
  the perceived physical value scale, and at the subdomain level, 4 subscales: the fitness, athletic competence, physical appearance and strength. It has 25 items
  * The subject responds on the Likert scale in 6 increasing degrees (it looks like me 1: not at all, 2: very little, 3: a little, 4: enough, 5: a lot, 6: quite).
  * The score ranges from 5 to 30 for each scale, total score is averaged.
Depression: Center for Epidemiologic Studies Depression Scale, CES-D | 1 year
  • The CES-D assesses the frequency and severity of depressive symptoms presented by the general population.
  The questionnaire has 20 items.
  * The subject indicates on a 4-point Likert scale ranging from "almost never" to "almost always", a frequency at which he usually feels the symptoms listed.
  * Score is calculated from 0 to 60 (maximum score indicating strong expression of symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No